CLINICAL TRIAL: NCT07249541
Title: Investigation of the Relationship Between Hypermobility, Foot Posture, and Scoliosis Severity in Adolescents With Idiopathic Scoliosis
Brief Title: Hypermobility, Foot Posture, and Scoliosis Severity
Acronym: AIS
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Tuğçe Yavuz, Principal Investigator, Istinye University
Other Study IDs: 25-121
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Joint Hypermobility; Adolescent Idiopathic Scoliosis; Foot Posture
MeSH Terms: conditions — Joint Instability | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescent Idiopathic Scoliosis Group: Participants diagnosed with Adolescent Idiopathic Scoliosis will undergo assessments of hypermobility (Beighton Score), foot posture (Foot Posture Index), and scoliosis severity (Cobb angle).
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Participants diagnosed with Adolescent Idiopathic Scoliosis will undergo assessments of hypermobility (Beighton Score), foot posture (Foot Posture Index), and scoliosis severity (Cobb angle).

SUMMARY:
Adolescent Idiopathic Scoliosis is a three-dimensional spinal deformity that may also affect joint mobility, lower limb alignment, and overall posture. Joint hypermobility and foot posture abnormalities, including pronation or supination, are commonly observed in adolescents and may contribute to postural imbalance or altered biomechanical loading. However, the relationship between hypermobility, foot posture, and the severity of scoliosis remains unclear.

The aim of this study is to examine whether generalized joint hypermobility and foot posture characteristics are associated with Cobb angle severity in adolescents diagnosed with Adolescent Idiopathic Scoliosis. Hypermobility will be assessed using the Beighton Score, and foot posture will be evaluated with the Foot Posture Index. Understanding these associations may help clinicians better evaluate biomechanical factors related to scoliosis and guide future preventive or therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Adolescent Idiopathic Scoliosis
* Age 10-19 years
* Cobb angle ≥ 10° on standing Anterior-Posterior radiograph
* Ability to participate in physical assessments
* Voluntary consent to participate

Exclusion Criteria:

* Neuromuscular, syndromic, or congenital scoliosis
* Previous spinal surgery
* Lower extremity orthopedic conditions affecting foot posture
* Neurological or rheumatological disorders affecting joint mobility
* Communication or cognitive difficulties limiting participate

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of adolescents aged 10 to 19 years who have been clinically and radiographically diagnosed with Adolescent Idiopathic Scoliosis. Participants must have a Cobb angle of at least 10° and be able to complete physical assessments, including hypermobility and foot posture evaluations.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Foot Posture Index-6 | 4 weeks
  The Foot Posture Index-6 is a reliable and valid clinical assessment tool used to objectively evaluate foot posture in the pronation-supination spectrum. The assessment is performed with the individual in a relaxed standing position and is based on six observational criteria. The total score ranges from -12 to +12, where higher scores indicate a more pronated foot posture, while lower scores reflect a more supinated posture. A score close to 0 represents a neutral foot posture.
The Beighton Test | 4 weeks
  This is a standardized and easily applicable clinical assessment method used to determine joint hypermobility. The total score for the nine-item test ranges from 0 to 9. A total score of ≥4 indicates the presence of hypermobility. It is scored out of 9 points; each positive finding is evaluated as 1 point.

SECONDARY OUTCOMES:
Feiss Line Test | 4 weeks
  Used to evaluate the structural characteristics of the arch of the foot. In this test, the position of the navicular tubercle above or below a line drawn by aligning the medial malleolus, navicular tubercle, and first metatarsal head indicates the presence of pes planus or pes cavus.
Sit-Reach Test | 4 weeks
  This is a common field test that evaluates the flexibility of the hamstring and lumbar muscles. The participant sits in a straight position, knees straight, and the soles of their feet touching the test box, reaching forward; the distance between their toes indicates the level of flexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No